CLINICAL TRIAL: NCT02714244
Title: Evaluation of the E/e' Ratio of the Mitral Annulus Measured by Transesophageal Echocardiography in Predicting Fluid Responsiveness.
Brief Title: Evaluation of the E/e' Ratio of the Mitral Annulus in Predicting Fluid Responsiveness.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Montreal Heart Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2014-1671
Record Dates: First submitted 2016-03-03; First posted 2016-03-21 (Estimated); Last update posted 2017-09-07 (Actual); Status verified 2016-12

CONDITIONS: Left Ventricular Function Diastolic Dysfunction; Fluid Responsiveness
MeSH Terms: interventions — Ringer's Lactate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Volume expansion — Volume expansion with rapid administration of 500 ml of crystalloid
  Other Names: Lactate Ringer

SUMMARY:
Diastolic function may be evaluated by different measurements on transesophageal echocardiography (TEE). They include mitral inflow velocities obtained by pulsed-wave doppler (PW) : peak early diastolic velocity (E) and late diastolic velocity (A). Mitral annulus velocities, early diastolic (e') and late diastolic (a') are obtained by tissue doppler imaging (TDI). The ratio E/e' reflects left ventricular filling pressure and, as such, might be a predictor of fluid responsiveness.

The aim of this study is to evaluate the predictive value of the mitral valve E/e' ratio for fluid responsiveness among patients undergoing coronary bypass graft surgery. Fluid responsiveness being defined as an increase in stroke volume of ≥ 15%.

After induction of anesthesia, patients will have their diastolic function evaluated by means of E/e' and other measures. They will then be administered an intravenous bolus of 500 mL of Lactate Ringer® along with passive leg raising (PLR). Stroke volume and fluid responsiveness will be assessed by the thermodilution method (Swan-Ganz catheter) and the FloTrac® device. Fluid responders will be compared to non-responders to evaluate the relationship between E/e' ratio and fluid responsiveness.

ELIGIBILITY:
Inclusion Criteria:

* Patients >18 yrs, undergoing elective coronary artery bypass grafting or surgery will be included.

Exclusion Criteria:

* Significant mitral valvular heart disease (mitral regurgitation ≥ 2/4 or stenosis)
* Significant right sided valvular heart disease (tricuspid regurgitation ≥ 2/4)
* Intracardiac shunts
* Emergency surgery
* Non-sinusal rythme
* Clinical evidence of decompensated heart failure
* Clinical evidence of decompensated pulmonary hypertension
* Renal insufficiency with creatinine clairance ≤ 30 cc/min or dialysis
* Contraindications to TEE, including esophageal disease or unstable cervical spine
* CVP ≥ 15 mm Hg or PCWP ≥ 18 mm Hg immediately before fluid infusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2016-01; Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Mitral valve E/e' ratio for prediction of fluid responsiveness | TEE images taken within the 15 minutes before fluid administration and responsiveness evaluation within the 5 minutes following fluid administration and leg raising
  TEE evaluation of mitral inflow velocities and mitral annulus velocities measured right before fluid administration as a predictor of fluid responsiveness defined as an increase of 15% or more of the stroke volume

SECONDARY OUTCOMES:
Pulmonary capillary wedge pressure (PCWP) a-wave to v-wave ratio of the for prediction of fluid responsiveness | Waveform measured within the 15 minutes preceding fluid administration and responsiveness evaluation within the 5 minutes following fluid administration and leg raising
  a-wave on v-wave ratio of the pulmonary capillary wedge pressure (PCWP) curve for prediction of fluid responsiveness defined as an increase of 15% or more of the stroke volume
Pulse pressure variation (PPV) for prediction of fluid responsiveness | PPV measured within the 15 minutes preceding fluid administration and responsiveness evaluation within the 5 minutes following fluid administration and leg raising
  Pulse pressure variation (PPV) measured on arterial pressure curve for prediction of fluid responsiveness defined as an increase of 15% or more of the stroke volume
Stroke volume variation (SVV) for prediction of fluid responsiveness | SVV measured within the 15 minutes preceding fluid administration and responsiveness evaluation within the 5 minutes following fluid administration and leg raising
  Stroke volume variation (SVV) directly measured by FloTrac/Vigileo® with its intrinsic algorithm for prediction of fluid responsiveness defined as an increase of 15% or more of the stroke volume

CONTACTS AND LOCATIONS:
Locations (1):
- Montreal Heart Institute, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Courbe A, Perrault-Hebert C, Ion I, Desjardins G, Fortier A, Denault A, Deschamps A, Couture P. Should we use diastolic function parameters to determine preload responsiveness in cardiac surgery? A pilot study. J Anesth Analg Crit Care. 2021 Oct 30;1(1):12. doi: 10.1186/s44158-021-00014-7. PMID 37386580